CLINICAL TRIAL: NCT03316144
Title: A Phase I Study of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of Recombinant Humanized Anti-PD-1 Monoclonal Antibody for Injection in Patients With Recurrent Malignant Lymphoma
Brief Title: Safety, Tolerability, Pharmacokinetics & Pharmacodynamics of Toripalimab for Patients With Recurrent Malignant Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Junshi-JS001-011
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Malignant Lymphoma
Keywords: immunotherapy; check point inhibitor; PD-1 antibody; phase 1 trial; Malignant Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 mg/kg Toripalimab (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 1mg/kg Q2w until disease progresses or unacceptable tolerability occurs
  Interventions: Biological: Toripalimab
- 3 mg/kg Toripalimab (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 3mg/kg Q2w until disease progresses or unacceptable tolerability occurs
  Interventions: Biological: Toripalimab
- 10 mg/kg Toripalimab (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 10mg/kg Q2w until disease progresses or unacceptable tolerability occurs
  Interventions: Biological: Toripalimab

INTERVENTIONS:
Biological: Toripalimab — Dose escalation study evaluating three dose levels (1, 3 and 10 mg/kg) of JS001. Subjects will be assigned to a dose schedule in the order of study entry.
  Other Names: JS001, TAB001

SUMMARY:
The primary objective is to assess the safety and tolerability of JS-001 in subjects with recurrent malignant lymphoma, and to evaluate its preliminary efficacy.

The secondary objectives are to: 1) characterize the single-dose and multi-dose pharmacokinetic (PK) profile of JS-001, 2) characterize the immunogenicity of JS-001; 3) assess the dose-efficacy relationship of JS-001 single agent, and 4) preliminarily evaluate biomarkers associated with the efficacy of JS-001.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign Informed Consent;
* Re-entry into the study is allowed with a second informed consent;
* Willing to provide blood sample for biomarker analysis(mandatory). The tissue sample is optional;
* A diagnosis of an advanced malignant tumor confirmed by histology or cytology (including typical Hodgkin's lymphoma and B cell source non-hodgkin's lymphoma);
* No standard of care for the patient;
* At least 1 measurable lesion;
* Aged 18-65 years;
* Anticipated life expectancy of at least 6 months;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* At least 4 weeks elapsed since receiving systemic chemotherapy;
* At least 4 weeks elapsed since receiving definite radiotherapy;
* At least 2 weeks since the last dose of systemic steroid therapy (>10 mg/day prednisone or equivalent);
* At least 4 weeks since receiving anti-cancer biotherapy;
* Recovered from previous treatment related adverse reaction; willing to use an acceptable contraceptive method;
* A negative pregnancy test for female subjects of childbearing potential;

Exclusion Criteria:

* Active central nervous system (CNS) metastases and/or carcinomatous meningitis;
* Known history of another primary solid tumor, unless the participant has undergone potentially curative therapy with no evidence of that disease for 2 years, or underwent successful definitive resection of basal or squamous cell carcinoma of the skin, or in situ cervical cancer;
* Active, known or suspected autoimmune disease.Autoimmune diseases caused by lymphoma are not included in this list;
* Patients who have had car-T cell therapy
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2,or anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4) blocking antibodies;
* Significant medical disease;
* Active infection;
* Active tuberculosis or history of tuberculosis with one year;
* Infection of Human immunodeficiency virus (HIV);
* A complication requiring immune-suppression;
* Received a live vaccine within 4 weeks prior to first dose of study drug pleural or abdominal effusion with symptoms;
* Drug or alcohol abuse (for subjects in the pharmacokinetic cohorts) ; evidence of interstitial lung disease;
* Active hepatitis B or C, or with significant risk of hepatitis reactivation;
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to monoclonal antibodies or drugs chemically related to the study drug. History of serious hypersensitivity reaction or serious hepatotoxicity related to any drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

SECONDARY OUTCOMES:
correlation analysis of PD-L1 expression of tumor | 6 months
Objective Response Rate (ORR) by irRC and RECIST 1.1 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Junyuan Qi, MD, PhD, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China